CLINICAL TRIAL: NCT07108998
Title: A Phase 2 Study of Epcoritamab as a Consolidation Therapy for 2nd Generation BTKi +/- Obinutuzumab in CLL/SLL Patients or Variants of This.
Brief Title: Study of Epcoritamab as a Consolidation Therapy in CLL/SLL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zulfa Omer (Other)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor-Investigator, Zulfa Omer, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-HEM-24-01; IST-EPCO-00035 (Other: Genmab)
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: CLL/SLL; CLL; SLL; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Small Lymphocytic Lymphoma Variant; Chronic Lymphocytic Leukemia Variants
Keywords: Epcoritamab; Obinutuzumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Epcoritamab + SOC (Experimental): Epcoritamab is the investigational product under study in combination with SOC drugs in this protocol. During C1, epcoritamab will be initiated using step-up dosing (SUD) C1D1 .16mg, C1D8 .8mg, C1D15 3 mg, C1D22 24 mg vs 48 mg (full dose) during safety lead in to determine the RP2D. On Cycles 2-3 the RP2D (24mg vs 48 mg) will be administered on Days 1, 8, 15, 22. Then Cycles 4-9 RP2D will be administered on Days 1 & 15. Then Cycle 10-12 RP2D on Day 1 of each cycle. Epcoritamab is administered subcutaneously. The SOC BTKi are oral medications administered daily during the trial period.
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Epcoritamab is the investigational product under study in combination with SOC drugs in this protocol. During C1, epcoritamab will be initiated using step-up dosing (SUD) C1D1 .16mg, C1D8 .8mg, C1D15 3 mg, C1D22 24 mg vs 48 mg (full dose) during safety lead in to determine the RP2D. On Cycles 2-3 the RP2D (24mg vs 48 mg) will be administered on Days 1, 8, 15, 22. Then Cycles 4-9 RP2D will be administered on Days 1 & 15. Then Cycle 10-12 RP2D on Day 1 of each cycle. Epcoritamab is administered subcutaneously. The SOC BTKi are oral medications administered daily during the trial period.

SUMMARY:
This is a phase 2 study of Epcoritamab as a consolidation therapy for 2nd generation BTKi +/- Obinutuzumab in CLL/SLL patients or patients with variants of this.

DETAILED DESCRIPTION:
This is a Phase II, multicenter trial, where we seek to test the hypothesis that administration of up to 12 cycles of epcoritamab following a 12 months or greater time period of acalabrutinib +/- obinutuzumab or zanubrutinib +/- obinutuzumab in patients who have attained a partial response or better will have a high CR conversion rate with uMRD that enables discontinuation of therapy and lead to durable remission. Additionally, Patients attaining this exceptional uMRD CR at completion of therapy will have evidence of autologous T-cell response toward the patient pre-treatment CLL cells. A safety lead in of the combination for the first 9 patients followed by Simon's 2 stage design will be implemented. Following our inclusion and exclusion criteria, eligible patients will be treated with subcutaneous epcoritamab for a total of 12 cycles while continuing their BTKi therapy. Patients will be assessed for disease response as defined by the iw-CLL 2018 response criteria following completion of cycle 6 and 12 of epcoritamab by peripheral blood labs, CT imaging and bone marrow biopsy for morphology and flow cytometry (if labs/imaging indicating CR) and MRD status through NGS assay (ClonoSEQ). MRD will be performed from bone marrow samples if BMBx is done, and if not done peripheral blood sample will be used for MRD status. All patients who complete 12 cycles of epcoritamab consolidative therapy will have the ability to continue BTKi as monotherapy regardless of MRD status, pending discussion with the patient and treating-physician.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of CLL or SLL meeting the established 2018 iwCLL diagnostic criteria or variant of CLL/SLL and has received a 2nd generation BTKi (acalabrutinib or zanubrutinib) +/- obinutuzumab for a minimum of 12 months as first line therapy.

   a) Note: Variation in flow cytometry is defined as patients who have atypical immunophenotyping for CLL (CD5 negative, CD23 negative or surface expression of CD79b that is bright ) but clinically behave like CLL (leukocytosis, lymphadenopathy and splenomegaly) and have the FISH/Cytogenetics translocations(del 13q, trisomy 12, Del11q) or genomic features (XPO1, NOTCH1, SF3B1, FBXW7, MYD88, BIRC3, TRAF3, NFKBIE, SAMHD1, POT1, HIST1H1E, CHD2, ZMYM3, EGR2 and others) that are suggestive of CLL.
2. Attainment of Partial Response or greater with a 2nd generation BTKi (acalabrutinib or zanubrutinib) +/- obinutuzumab but detectable disease in blood or bone marrow by NGS ClonoSEQ.
3. Age ≥18 years.
4. ECOG performance status ≤2 (or Karnofsky ≥60%, see Appendix D).
5. Patients must have adequate organ and marrow function as defined below:

   Absolute neutrophil count ≥1,000/mcL, unless if neutropenia is due to underlying CLL bone marrow disease.

   Hemoglobin ≥8 g/dl unless if related to underlying CLL Platelets ≥50,000/ µL unless if related to underlying CLL Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (excepting Gilbert's syndrome, who may have a bilirubin > 1.5 × ULN, per discussion between the Investigator and the UC PI).

   AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN Glomerular filtration rate (GFR) Calculated GFR using CKD-EPI formula ≥ 30 (See Appendix E) or multiplying the estimate of GFR by an individual body surface area calculated using an appropriate formula and dividing by 1.73 m2.
6. Women of childbearing potential and non-sterile males must practice at least 1 of the following methods of birth control with their partner(s) throughout the study and for 4 months after discontinuing study drug:

   1. Total abstinence from sexual intercourse as the preferred lifestyle of the patient; periodic abstinence is not acceptable.
   2. Surgically sterile partner(s) by vasectomy, bilateral orchiectomy, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
   3. Intrauterine device.
   4. Hormonal contraceptives (oral, parenteral, vaginal ring or transdermal) for at least 1-month prior to study drug administration.
7. Women of childbearing potential must have a negative pregnancy result as follows: At Screening on a serum sample obtained within 7 days prior to the first study drug administration. If a urine pregnancy test at any timepoint during the study is positive or indeterminate, a serum pregnancy test will be performed for confirmation.
8. Non-sterile males must refrain from sperm donation, from initial study drug administration until 4 months after the last dose of study drug.
9. Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

1. Obtaining a CR or nodal PR with no detectable disease in blood or bone marrow after treatment with a 2nd generation BTKi (acalabrutinib or zanubrutinib) +/- obinutuzumab as assessed by Adaptive's NGS ClonoSEQ.
2. Absence of CD20 expression on CLL cells at pre-treatment.
3. Received any prior treatment ever with a CD3×CD20 bispecific antibody.
4. Organ transplant recipients are excluded except those with no active graft versus host disease (GVHD) requiring treatment within 12 months of beginning treatment on study.
5. Receipt of a live vaccine within 28 days prior to study treatment initiation.
6. Autoimmune diseases requiring high dose immunosuppressives (e.g., above 20 mg prednisone daily).
7. Central nervous system (CNS) disease(s) unless in the opinion of the investigator these would not preclude the patient from participation.
8. Known hypersensitivity to any of the components of the treatment drugs (see Investigators Brochure for a list of components).
9. Patients with active Richter's transformation.

   a. Note: the following will be eligible and not excluded: patients with accelerated phase or prolymphocytic progression
10. Patients who have received prior radiation therapy (RT) unless in the opinion of the investigator the prior receipt of RT will not adversely impact the patient's ability to participate.
11. Patients who require anti-coagulation with warfarin or equivalent Vitamin K antagonist.
12. Major surgery within 14 days prior to the first dose of study drug.
13. Patient has significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 180 days prior to the first dose of study drug, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification or left ventricular ejection fraction ≤ 40%.
14. Pregnant women, those planning to become pregnant during the study, and/or breastfeeding women are ineligible for participation.
15. Patient exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

    1. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds). No new IV therapy or intravenous antibiotics may be initiated within 2 weeks prior to first dose of study drug.
    2. Known poorly controlled human immunodeficiency virus (HIV) or active hepatitis B or C infection (active hepatitis B defined as HBsAg positive, or HBcAb positive with detectable HBV DNA load; active hepatitis C defined as HCV antibody positive with HCV RNA positive)
    3. Unexplained fever > 38.3°C within 7 days prior to the first dose of study drug administration (if the fever is considered attributed to the patient's malignancy or an explained infection, the Patient may be enrolled at the discretion of the Investigator).
16. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
uMRD CR as defined by negative leukemia cells to the 10^6 | Post 12 cycles (approximately 336 days after the start of first cycle) of consolidative therapy with epcoritamab
  uMRD CR as defined by negative leukemia cells to the 10^6 after 12 cycles of consolidative therapy with epcoritamab measured by Adaptive's NGS MRD assay (ClonoSEQ) in patients who have attained a partial response or better with detectable disease after acalabrutinib or zanubrutinib +/- obinutuzumab treatment for a minimum of 12 cycles of therapy

SECONDARY OUTCOMES:
Safety measured by CTCAE v. 5. | Day 1 of Cycle 1 to 60 days after end of C12D28 (i.e., approximately 396 days after the start of intervention)
  Safety of epcoritamab given together with acalabrutinib or zanubrutinib in patients with CLL/SLL reported as frequency and severity of adverse events using CTCAE v. 5.
uMRD CR defined by negative leukemia cells to the 10^6 using NGG ClonoSEQ | Post 6 cycles (approximately 196 days after start of intervention) of consolidation with epcoritamab.
  uMRD CR defined by negative leukemia cells to the 10^6 using NGG ClonoSEQ after 6 cycles of consolidation with epcoritamab.
T-cell subsets levels measured by flow-cytometry | Baseline, pre-treatment on Cycle1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 7 Day 1 and end of Cycle 12. Each cycle is 28 days.
  T-cell subsets levels (include T-regulatory cells, TH17 T-cells, effector memory T-cells, central memory T-cells, naïve T-cells, and cytotoxic T-cells) at baseline, Day 1, Day 8, C2D1, C4D1, C7D1 and C12 D28 of consolidation with epcoritamab.
PFS defined as the interval between the first treatment day to the first sign of disease progression or death from any cause of patient | Post 12 cycles of consolidative epcoritamab (approximately 364 days from start of intervention).. Each cycle is 28 days.
  PFS defined as the interval between the first treatment day to the first sign of disease progression or death from any cause after receiving 12 cycles of consolidative epcoritamab.
OS defined as time from starting treatment until death of patients | Post 12 cycles of consolidative epcoritamab (approximately 364 days from start of intervention).. Each cycle is 28 days.
  OS defined as time from starting treatment until death of patients after receiving 12 cycles of consolidative epcoritamab.

OTHER OUTCOMES:
T-cell cytotoxicity against primary pretreatment CLL cells | Baseline, Day 1, Day 8, Day 29 of Cycle 1, end of Cycle 3, Cycle 6 and Cycle 12 of consolidation with epcoritamab. Each cycle is 28 days.
  T-cell cytotoxicity against primary pretreatment CLL identified by INF-gamma production in presence of ex-vivo incubated CLL cells at baseline, Day 1, Day 8, Day 29 of Cycle 1, end of Cycle 3, Cycle 6 and Cycle 12 of consolidation with epcoritamab.
T-cell proliferation against primary pretreatment CLL cells | Baseline, Day 1, Day 8, Day 29 of Cycle 1, end of Cycle 3, Cycle 6 and Cycle 12 of consolidation with epcoritamab. Each cycle is 28 days.
  T-cell proliferation against primary pretreatment CLL cells through identifying different T cell cells receptor(TCR) using next generation sequencing at baseline, Day 1, Day 8, Day 29 of Cycle 1, end of Cycle 3, Cycle 6 and Cycle 12 of consolidation with epcoritamab.
Cytokine production against autologous CLL cells | Baseline, Day 1, Day 8, Day 29 of Cycle 1, end of Cycle 3, Cycle 6 and Cycle 12 of consolidation with epcoritamab. Each cycle is 28 days.
  Cytokine levels ( e.g. IL-6, TNF-alpha) produced using flow cytometry against CLL cells at baseline, Day 1, Day 8, Day 29 of Cycle 1, end of Cycle 3, Cycle 6 and Cycle 12 of consolidation with epcoritamab.
Tumor features of patients who respond to epcoritamab therapy and then relapse following receipt of this treatment. | Screening, Baseline pre-treatment on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 7 Day 1, end of Cycle 12 (or at EOT) and Relapse. Each cycle is 28 days.
  To determine pre-treatment and serial tumor features changes including development of new mutations and change in genomics through whole exon sequencing and single cell sequecning that are associated with response in CLL patients receiving epcoritamab at the following timepoints Screening, Baseline pre-treatment on C1D1, C1D8, C2D1, C4D1, C7D1, end of C12 (or at EOT) and Relapse.
Pre-treatment and serial findings associated with CRS in CLL patients receiving epcoritamab. | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 7 Day 1, end of Cycle 12. Each cycle is 28 days.
  To determine pre-treatment and serial levels of ferritin, soluble CD163 , IL-6, IFN-gamma through flow-cytometry that are associated with CRS in CLL patients receiving epcoritamab through measurement of INF gamma production.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided